CLINICAL TRIAL: NCT07358403
Title: Clinical Instrumental Evaluation of the Efficacy of a Dietary Supplement Claiming Anti Hair Loss Properties
Brief Title: Evaluation of the Dietary Supplement Efficacy Against Hair Loss in Subjects Suffering From Hair Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lacer S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IT0006736/24
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Androgenetic Alopecia (AGA); Chronic Telogen Effluvium
MeSH Terms: conditions — Alopecia | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dietary supplement capsule (Experimental): Dietary supplement capsule was taken by the subjects daily during 6 months
  Interventions: Dietary Supplement: Dietary supplement capsule use for hair loss
- Dietary supplement capsule placebo (Placebo Comparator): Dietary supplement capsule placebo was taken by the subjects daily during 6 months
  Interventions: Dietary Supplement: Dietary supplement capsule placebo use for hair loss
- Dietary supplement drinkable (Experimental): Dietary supplement drinkable was taken by the subjects daily during 6 months
  Interventions: Dietary Supplement: Dietary supplement drinklable use for hair loss
- Dietary supplement drinkable placebo (Placebo Comparator): Dietary supplement drinkable placebo was taken by the subjects daily during 6 months
  Interventions: Dietary Supplement: Dietary supplement drinklable placebo

INTERVENTIONS:
Dietary Supplement: Dietary supplement capsule use for hair loss — Dietary supplement capsule use for hair loss, once a day during 6 months.
  Arms: Dietary supplement capsule
Dietary Supplement: Dietary supplement capsule placebo use for hair loss — Dietary supplement capsule placebo use for hair loss, once a day during 6 months.
  Arms: Dietary supplement capsule placebo
Dietary Supplement: Dietary supplement drinklable use for hair loss — Dietary supplement drinklable use for hair loss, once a day during 6 months.
  Arms: Dietary supplement drinkable
Dietary Supplement: Dietary supplement drinklable placebo — Dietary supplement drinklable placebo use for hair loss, once a day during 6 months.
  Arms: Dietary supplement drinkable placebo

SUMMARY:
The goal of this study was to learn if dietary supplement in capsules and drinkable works to help hair loss in volunteers with chronic telogen effluvium and androgenetic alopecia and learn about its safety. The main questions it aims to answer are:

* Does dietary supplement in capsules and drinkable reduces hair loss in women and men suffering from chronic telogen effluvium or androgenetic alopecia?
* Were the products well accepted by the subjects from their´s perspective? Researchers will compare dietary supplement in capsules and drinkable to a placebo (a look-alike substance that contains no active ingredients) to see if dietary supplements works to reduce hair loss.

Participants will:

* Take assigned diatry supplement in capsule or drinkable or a placebo every day for 6 months
* Visit the study facility once every 3 months for evaulations
* Keep a diary of the product use

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male subjects, including at least 70% female subjects aged over 30 years old ✓ Caucasian ethnicity
* Aged between 18 and 62 years old (extreme included)
* 50% of subjects with chronic telogen effluvium (stage from 2 to 4, according to Sinclair scale for female pattern hair loss in women and modified Sinclair scale for female pattern hair loss in men)
* 50% of subjects with androgenetic alopecia (AGA): female subjects Ludwig scale (score I-II) and male subjects Hamilton- Norwood scale (vertex II-III)
* Subjects aware of the study procedures and having signed an informed consent form
* Subjects registered with National Health Service (NHS)
* Subjects certifying the truthfulness of the personal data disclosed to the investigator
* Subjects able to understand the language used in the investigation and to respect the instructions given by the investigator as well as able to respect the study constraints and specific requirements
* The pharmacological therapy (except for the pharmacological therapy in the non-inclusion criteria) should be stable for at least one month without any changes expected or planned during the study
* Commitment not to change the daily routine or the lifestyle
* Subject informed about the study procedures and having signed the privacy policy

Exclusion Criteria:

* Subjects who do not fit the inclusion criteria.
* Subjects with acute or chronic diseases able to interfere with the outcome of the study or that are considered dangerous for the subject or incompatible with the study requirements
* Subjects participating or planning to participate in other clinical trials
* Subjects deprived of freedom by administrative or legal decision or under guardianship
* Subjects not able to be contacted in case of emergency
* Subjects admitted to a health or social facility
* Subjects planning a hospitalization during the study
* Subjects who participated in a similar study without respecting an adequate washout period (3 months)
* Alimentary/Eating disorders (i.e., bulimia, psychogenic eating disorders, etc.)
* Food allergy or food intolerances
* Impaired immune system due to i-mmunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications
* Subjects who have any type of gastrointestinal disease or disorders (Chrons disease, colitis, irritable bowel syndrome, intestinal malabsorption)
* Pharmacological treatment (topic or systemic) known to interfere with the tested product or having effect on metabolism (e.g.: anticoagulants, antidepressants, drugs used to lower cholesterol levels, antiviral drugs and beta-blockers)
* Subjects having frequent stomach burn
* Cosmetic treatment known to interfere with the tested product (e.g.: anti-hair loss shampoo, antihair loss food supplements, anti-hair loss serum) during the study and in the last 3 months before study start
* Subjects who intends to carry out any straightening, permanent or other treatments on hair (hair botox,etc)
* Subjects with drandruff, seborrheic dermatitis or any other hair condition
* Subjects having a skin disease or condition liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* Subjects that have shown allergies or sensitivity to cosmetic products, drugs, patch or medical devices
* Subject breastfeeding, pregnant or not willing to take necessary precautions to avoid pregnancy during the study (for the women of childbearing potential)

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the hair density at 3 and 6 months | From the baseline, at 3 months and at the end of the study (6 months).
  Pictures of chosen area of the scalp are taken and the number of hairs per cm2 is counted.

SECONDARY OUTCOMES:
Assessment of product acceptability and perceived efficacy at 3 and 6 months | On 3 months and 6 months of product use.
  Subjects responded questionnaire regarding product cosmetic qualities and efficacy where percentage of agreement with the statement was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Complife Italia, San Martino Siccomario, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
The results will be shared in the paper.

DOCUMENTS (1):
  • Study Protocol (2024-12-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT07358403/Prot_000.pdf